CLINICAL TRIAL: NCT06982352
Title: Phase 1b Randomized, Double Blind, Placebo-controlled Study to Evaluate Safety, Tolerability and Pharmacokinetics of LPX-TI641 in Patients With Atopic Dermatitis and Psoriasis
Brief Title: Safety and Pharmacokinetics of LPX-TI641 in Atopic Dermatitis and Psoriasis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LAPIX Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LPX641-103
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis (AD); Psoriasis (PsO)
Keywords: phase 1 study; safety; pharmacokinetics
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis

STUDY DESIGN:
Intervention Model Description: This is a Phase 1b, multi-center, randomized, double-blind, parallel-group, placebo-controlled multiple ascending doses (MAD) study in participants with atopic dermatitis, or psoriasis.
  There will be 2 cohorts, one for each indication. Each cohort will consist of ~12-24 participants (Total ~up to 48 participants). . Each cohort will consist of ~20-to-24 participants (Total ~up to 48 participants in the trial) treated QD for 28 days.
  The first cohort is for Atopic Dermatitis (AD), where the participants will receive 150 mg LPX-TI641 QD or placebo for 28 days (3:1, treatment: placebo randomization).
  The Plaque psoriasis (PsO) cohort may be treated concurrently or sequentially with the Atopic Dermatitis (AD) cohort. Participants in the PsO cohort will be randomized in a 3:1 ratio for LPX-TI641 150 mg QD: placebo QD treatment for 28 days.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psoriasis (Experimental): LPX-TI641 or Placebo
  Interventions: Drug: LPX-TI641; Drug: Placebo
- Atopic dermatitis (Experimental): LPX-TI641 or Placebo
  Interventions: Drug: LPX-TI641; Drug: Placebo

INTERVENTIONS:
Drug: LPX-TI641 — Oral administration QD for 28 consecutive days
Drug: Placebo — Placebo an identical oral formulation without the LPX-TI641.

SUMMARY:
The goal of this clinical trial is to study the drug LPX-TI641 in patients with atopic dermatitis and psoriasis. We will compare the safety and tolerability of LPX-TI641 to placebo ( a look-alike solution) that contains no drug. We will also evaluate the plasma pharmacokinetics of LPX-TI641. LPX-TI641 (or placebo) will be administered orally for 28 days.

DETAILED DESCRIPTION:
This is a Phase 1b, multi-center, randomized, double-blind, parallel-group, placebo-controlled multiple dose study in participants with atopic dermatitis or psoriasis.

There will be 2 cohorts, one for each indication. Each cohort will consist of ~ 16-24participants (Total ~up to 48 participants).

The Primary objective of the study is to evaluate the safety and tolerability after multiple oral doses of LPX-TI641 in participants with AD and PsO.

And the secondary objective of the study is to evaluate the plasma pharmacokinetics after multiple oral doses of LPX-TI641 in participants with AD and PsO.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed an Informed Consent Form (ICF) prior to any study-specific procedures being performed
2. ≥ 18 years old, irrespective of their race and ethnicity.
3. Body Mass Index (BMI) 18.0-40.0 kg/m2, inclusive, at screening.
4. Participants are willing and able to adhere to study protocol requirements and restrictions including but not limited to scheduled outpatient visits, inpatient stay, laboratory tests, and 12-lead ECGs.
5. The subject must be judged to be in good health by the investigator to participate in the study, based on clinical evaluations, including laboratory safety tests, medical history, physical examination, vital signs and 12-lead ECG completed at the screening visit and prior to the first dose of study drug.
6. Female subject is postmenopausal (at least 1 year; to be confirmed by FSH if less than 2 years since last menstrual period), permanently sterilized (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy) or if of childbearing potential and engaged in sexual activity that can result in pregnancy must agree to use any two of the highly effective contraception methods listed below. Male participants with a partner of childbearing potential must also agree to use any two of the highly effective contraception methods listed below between them and their partner. This criterion must be followed from screening visit to 6 weeks after the last dose in females and for 90 days after the last dose for males.

   The following applies to all female participants with childbearing potential and female partners of male participants enrolled in the study.
   1. Implantable progestogen-only hormone contraception associated with inhibition of ovulation.
   2. Intrauterine device.
   3. Intrauterine hormone-releasing system.
   4. Bilateral tubal occlusion.
   5. Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation:
   6. Oral
   7. Intravaginal
   8. Transdermal
   9. Injectable
   10. Progestogen-only hormone contraception (oral or injectable) associated with inhibition of ovulation.
   11. Vasectomized partner
   12. Sexual abstinence -this is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated about the duration of the study and the preferred and usual lifestyle of the participant.
   13. A combination of male condoms with either cervical cap, diaphragm, or sponge with spermicide (double-barrier methods)

       The following applies to all male participants in the study:
   14. Sexual abstinence- this is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence must be evaluated for the study and the participant's preferred and usual lifestyle.
   15. A combination of male condoms with either cervical cap, diaphragm, or sponge with spermicide (double-barrier methods).
   16. Vasectomy
7. Negative serum B-human chorionic gonadotropin test at screening (for all females) and negative urine pregnancy at randomization (Day 1) (females of childbearing potential) prior to administration of investigational product.

   For Atopic Dermatitis Cohort:
8. Diagnosis of AD at least 12 months prior to screening, as defined by the American Academy of Dermatology: Guidelines of care for the management of atopic dermatitis (Eichenfield 2014):

   1. EASI score ≥ 16 at Screening and baseline (Day 0)
   2. vIGA score of ≥3 at screening and baseline (Day 0)
   3. ≥10% of body surface area (BSA) involvement at screening and baseline (Day 0)
   4. Peak pruritis NRS≥4 (average score of daily scores 7 days before Day 0)
9. History, documented by a physician and/or investigator, of inadequate response to existing topical medications within 6 months preceding screening, or history of intolerance to topical therapy as defined by at least 1 of the following:

   1. Inability to achieve good disease control defined as mild disease or better (e.g., IGA≤2) after use of at least a medium potency topical corticosteroid (TCS) for at least 4 weeks, or for the maximum duration recommended by the product prescribing information (e.g. 14 days for super potent TCS), whichever is shorter (Note: a TCS may be used with or without topical calcineurin inhibitors [TCNIs])
   2. Documented history of clinically significant adverse reactions with the use of TCS, such as skin atrophy, allergic reactions, or systemic effects that, in the opinion of the investigator, outweigh the benefits of retreatment
   3. Failed systemic therapies intended to treat AD within 6 months preceding screening (will be considered as having inadequate response to topical therapy)
10. Documented history of clinically significant adverse reactions with the use of TCS, such as skin atrophy, allergic reactions, or systemic effects that, in the opinion of the investigator, outweigh the benefits of retreatment

    For Plaque Psoriasis Cohort:
11. Confirmed diagnosis of plaque psoriasis for at least 6 months prior to baseline (Day 0)
12. Plaque psoriasis involving ≥10% body surface area (BSA) in the affected skin other than the face and scalp at screening and baseline (Day 0)
13. Static Physician's Global Assessment (sPGA) score ≥3 at screening and baseline (Day 0)
14. PASI score of ≥12 at screening and baseline (Day 0)
15. Subject must be candidate for phototherapy or systemic therapy
16. Subject had no significant flare in psoriasis for at least 3 months before screening

Exclusion Criteria:

1. History of clinically significant medical conditions or any other reason that in the opinion of the PI would interfere with subject's participation in this study
2. History of clinically significant drug or alcohol abuse per the PI's opinion within the last 6 months.
3. Pregnant or lactating women or women currently undergoing infertility treatments or women who intend to become pregnant during the time of study or for 6 weeks after last dose.
4. Presence of skin comorbidities that would interfere with study assessment or response to treatment
5. Any known history of malignancy within 5 years other than completely treated non-metastatic basal cell carcinomas or squamous cell carcinomas of the skin or localized carcinoma in situ of the cervix.
6. Patients who are currently experiencing a skin infection that requires treatment, or is currently being treated, with topical or systemic antibiotics
7. Symptomatic herpes zoster within 3 months of screening
8. For the plaque psoriasis cohort,

   1. Unstable forms of PsO (acute guttate PsO, psoriatic erythroderma, generalized pustular PsO, or other unstable form as judged by the investigator), or drug-induced psoriasis.
   2. History of any non-PsO disease that required treatment with oral or parenteral corticosteroids for more than 2 weeks within the past 24 weeks prior to signing the informed consent form (ICF)
9. Receipt of an investigational therapy less than 3 months or 5 drug-elimination half-lives (whichever is longer) prior to first administration of study treatment and during the study
10. Use of the following topical medications/emollients which could affect assessment of disease activity for at least 2 weeks prior to baseline (Day 0) and throughout the study:

    1. Topical corticosteroids or topical immune modulators (e.g. tacrolimus or pimecrolimus)
    2. Topical phosphodiesterase type 4 (PDE 4) inhibitor or JAK inhibitors or aryl hydrocarbon receptor agonists
    3. Topical or systemic antihistamines
    4. Use of emollients.
11. Receipt of any of the following excluded therapies as per below and throughout the study:

    1. Oral retinoids within 2 weeks of Day 0
    2. Systemic immunosuppressive/immunomodulating therapy (such as but not limited to systemic glucocorticoids, cyclosporine, mycophenolate mofetil, methotrexate, azathioprine, apremilast, or oral JAK inhibiting agents or phototherapy within 4 weeks before screening visit. Stable dose of max 1200ug inhaled budesonide (or equivalent) is allowed.
    3. Any cell depleting therapy, anti-CD4, anti-CD5, anti-CD3 other than anti-CD20 such as rituximab, ocrelizumab, and ofatumumab. Patients who have received rituximab or other selective B lymphocyte depleting agents (including experimental agents) are eligible if they have not received such therapy for at least 1 year prior to screening
12. Biologics dugs including, but not limited to dupilumab, tralokinumab, ustekinumab, secukinumab, ixikizumab, anti-TNF inhibitors within 8 weeks or 5 drug elimination half-lives whichever is longer and throughout the study
13. Failed biologics due to efficacy including, but not limited to dupilumab, tralokinumab, ustekinumab, secukinumab, ixikizumab, anti-TNF inhibitors
14. PUVA or UVB phototherapy within 4 weeks prior to Day 0 and throughout the study.
15. Subject has clinical or laboratory evidence of active or latent tuberculosis (TB) infection at screening as assessed by QuantiFERON-TB-Gold or a purified protein derivative skin test or equivalent (or both if required per local guidelines) and chest X-ray. Chest X-rays taken within 2 months prior to screening may be used instead of during screening if there is documentation showing no evidence of infection or malignancy as read by qualified physician.
16. Any active or recurrent infection within 1) the past 8 weeks prior to screening requiring IV/hospitalization or 2) the past 2 weeks prior to screening requiring oral antibiotics.
17. Laboratory values of the following at the Screening Visit:

    1. Hemoglobin < 11 g/dL
    2. WBC <3.5X109/L
    3. Absolute neutrophil count (ANC) < 1500 cells/µL, (or < 1200 cells/µL for participants of African descent who are black)
    4. Aspartate aminotransferase or alanine aminotransferase > 2.0 x the upper limit of normal (ULN) or bilirubin >= ULN;
    5. Bilirubin > ULN
    6. Platelets < 100,000 cells/[mm^3] (10^9/L)
    7. Clinically significant abnormal screening laboratory results as evaluated by the Investigator
18. Acutely worsened renal function within past 3 months prior to screening or estimated GFR by CDK-EPI creatinine equation with adjustment for body surface area <60ml/min.
19. Subject has any clinically significant finding on 12-lead ECG at screening or admission. NOTE: QTc(F) interval of >450 msec in male participants or >470 msec in female participants will be the basis for exclusion from the study. ECG may be repeated once for confirmatory purposes if initial values obtained exceed the limits specified.
20. Subject with positive results for HBsAg (hepatitis B surface antigens) and/or HBcAb (Hepatitis B core antibodies) and/or HCV Ab (hepatitis C antibodies) confirmed by HCV RNA, and/or HIV Ab (human immunodeficiency virus antibodies).
21. Blood loss of >250 mL or donated blood within 56 days or donated plasma within 7 days of screening.
22. Recent vaccination with live attenuated vaccines such as influenza, MMR, Herpes zoster, varicella, yellow fever, Rotavirus vaccine, etc., or inactivated vaccines such as Hepatitis A, rabies vaccine, etc. 30 days prior to screening visit
23. Subject has known sensitivity to any of the components of the investigational product.
24. Subject is investigative site personnel, sponsor personnel, or a member of their immediate families (spouse, parent, child or sibling whether biological or legally adopted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability after multiple oral doses of LPX-TI641 in participants with PsO and AD. | 84 days
  Rate and severity of treatment-emergent adverse events, including serious adverse events.

SECONDARY OUTCOMES:
To evaluate the plasma pharmacokinetics after multiple oral doses of LPX TI641 in participants with PsO and AD. | 24 hours on Day 1 and 24 hours on Day 28
  Measure Area Under the Concentration Time Curve after single dose and at Steady State

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Red River Research Partners, Fargo, North Dakota
  - Clinical Investigations of Texas, Dallas, Texas
- Triumpharma Clinical Research Unit at AlEssra Hospital, Amman, Jordan, Jordan